CLINICAL TRIAL: NCT04641507
Title: Comparative Study Between Tadalafil Versus Tamsulosin as a Medical Expulsive Therapy for Lower Ureteric Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Saleh Mostafa, Urology specialist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/30042019/Saleh
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Lower Ureteric Stones

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin treated group (Active Comparator): 83 patient with lower ureteric stone will take tamsulosin 0.4 mg once daily .Therapy will be given for a maximum of 4 weeks.
  Interventions: Drug: Tadalafil versus tamsulosin as MET
- Tadalafil treated group (Active Comparator): 83 patients with lower ureteric stone will take tadalafil 10 mg once daily. Therapy will be given for a maximum of 4 weeks.
  Interventions: Drug: Tadalafil versus tamsulosin as MET

INTERVENTIONS:
Drug: Tadalafil versus tamsulosin as MET — 166 patients with lower ureteric stone will be randomaized using computer-based randomization charts equally into 83 patients (Group A) treatment with tamsulosin 0.4 mg once daily or 83 patients (Group B) treatment with tadalafil 10 mg once daily. Therapy will be given for a maximum of 4 weeks.

SUMMARY:
The aim of the work is to compare the efficacy of tadalafil and tamsulosin as a medical expulsive therapy for lower ureteric stones

DETAILED DESCRIPTION:
Gradually increasing incidence rate of kidney stone is a significant concern of medical world. Genetics and/or life style accelerate the kidney stone formation (Urolithiasis). Sometimes, it is stuck up in ureter especially distal ureter; hence called as lower ureteral stone (LUS) and causes intense flank pain beside urinary obstruction.

The ureter contains α adrenergic receptors along its entire length with the highest concentration in the distal ureter.

There has been a steep rise in minimally invasive procedures but medical expulsive therapy (MET) is still regarded as an established treatment option for the management of distal ureteric stones.

Stone location, size, number, ureteric spasm, mucosal oedema or inflammation, and ureteric anatomy are the factors affecting passage of ureteric stones.

Drugs that expel stones might act by relaxing ureteral smooth muscle through inhibition of calcium channel pumps or α-1 receptor blockade. Tamsulosin is one of the most commonly used α-blockers.

Phosphodiesterase inhibitors (PDEi) are a class of drugs that inhibit the breakdown of cAMP and cGMP, enhancing smooth muscle relaxation. Therefore, PDEi may be able to decrease ureteral spasm and facilitate stone passage. Tadalafil is a selective PDE5i and because of its smooth muscle relaxation property, tadalafil received the US Food and Drug Administration approval for lower urinary tract symptoms with benign prostatic hyperplasia and erectile dysfunction.

Monotherapy with tadalafil or tamsulosin similarly improved lower urinary tract symptoms had already been demonstrated .

With demonstration of in vitro effects of phosphodiesterase-5 inhibitor (PDE5i) as tadalafil on isolated human ureteral smooth muscle, interest in use of PDE5i as MET has increased.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patient have a distal ureteric stone of 5-9 mm in greatest dimension
* Patient diagnosed by ultrasonography of the kidney, ureter, and bladder , X-ray KUB and noncontrast computed tomography scan.

Exclusion Criteria:

* Pregnant or lactating mothers.
* Patients have UTI.
* Patients have severe hydroureteronephrosis.
* Patients have multiple ureteric stones.
* Patients have solitary kidney.
* Patients have acute or chronic renal failure.
* Patients have previous therapies for the stone.
* Patients with history of open surgery/endoscopic interventions.
* Patients have ureteric strictures.
* Patients take concomitant treatment with calcium antagonists, β-blockers, corticosteroids or nitrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-05 (Estimated)

PRIMARY OUTCOMES:
Lower ureteric stone expulsion | 4 weeks
  Measuring lower ureteric stone expulsion rate with tadalafil versus tamsulosin

CONTACTS AND LOCATIONS:
Overall Officials: Amr Masoud, Doctorate, Study Chair — Head of urology department
Locations (1):
- Ahmed Saleh, Giza, Egypt

REFERENCES:
- [Background] Gratzke C, Uckert S, Kedia G, Reich O, Schlenker B, Seitz M, Becker AJ, Stief CG. In vitro effects of PDE5 inhibitors sildenafil, vardenafil and tadalafil on isolated human ureteral smooth muscle: a basic research approach. Urol Res. 2007 Feb;35(1):49-54. doi: 10.1007/s00240-006-0073-1. Epub 2006 Nov 11. PMID 17102958
- [Background] Oelke M, Giuliano F, Mirone V, Xu L, Cox D, Viktrup L. Monotherapy with tadalafil or tamsulosin similarly improved lower urinary tract symptoms suggestive of benign prostatic hyperplasia in an international, randomised, parallel, placebo-controlled clinical trial. Eur Urol. 2012 May;61(5):917-25. doi: 10.1016/j.eururo.2012.01.013. Epub 2012 Jan 20. PMID 22297243
- [Background] Pietropaolo A, Proietti S, Geraghty R, Skolarikos A, Papatsoris A, Liatsikos E, Somani BK. Trends of 'urolithiasis: interventions, simulation, and laser technology' over the last 16 years (2000-2015) as published in the literature (PubMed): a systematic review from European section of Uro-technology (ESUT). World J Urol. 2017 Nov;35(11):1651-1658. doi: 10.1007/s00345-017-2055-z. Epub 2017 Jun 7. PMID 28593477
- [Background] Seitz C, Liatsikos E, Porpiglia F, Tiselius HG, Zwergel U. Medical therapy to facilitate the passage of stones: what is the evidence? Eur Urol. 2009 Sep;56(3):455-71. doi: 10.1016/j.eururo.2009.06.012. Epub 2009 Jun 21. PMID 19560860
- [Background] Shabsigh R, Seftel AD, Rosen RC, Porst H, Ahuja S, Deeley MC, Garcia CS, Giuliano F. Review of time of onset and duration of clinical efficacy of phosphodiesterase type 5 inhibitors in treatment of erectile dysfunction. Urology. 2006 Oct;68(4):689-96. doi: 10.1016/j.urology.2006.05.009. No abstract available. PMID 17070333
- [Background] Tasian GE, Kabarriti AE, Kalmus A, Furth SL. Kidney Stone Recurrence among Children and Adolescents. J Urol. 2017 Jan;197(1):246-252. doi: 10.1016/j.juro.2016.07.090. Epub 2016 Aug 10. PMID 27521691